CLINICAL TRIAL: NCT03227354
Title: Open Study on the Validation of Non-invasive Absolute Intracranial Pressure Monitoring in Patients After Traumatic Brain Injury and Subarachnoid Hemorrhage
Brief Title: Validation of Non-invasive Absolute Intracranial Pressure Monitoring
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kienzler Jenny (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor-Investigator, Kienzler Jenny, Principal Investigator, Kantonsspital Aarau
Organization: Kantonsspital Aarau (Other)
Other Study IDs: aICP Validation 2
Record Dates: First submitted 2017-07-20; First posted 2017-07-24 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Intracranial Pressure Increase; Traumatic Brain Injury
Keywords: Medical Device
MeSH Terms: conditions — Intracranial Hypertension; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Vittamed 205 — non-invasive Intracranial Pressure measurement

SUMMARY:
Primary objective of this study is to assess the accuracy and precision of intracranial pressure (ICP) measurement in patients after traumatic brain injury and subarachnoid hemorrhage when using simultaneous, non-invasive measurement compared to standard, invasive, measurement.

Secondary objective: is to assess the correlation of intracranial pressure (ICP) measurement in patients after traumatic brain injury and subarachnoid hemorrhage between simultaneous, non-invasive measurement and standard, invasive,measurement

DETAILED DESCRIPTION:
Currently, ICP (Intracranial Pressure) can be measured only using invasive techniques. In a previous (pilot study) a non-invasive technique for measurement of ICP was investigated (based on simultaneously measuring of ophthalmic artery (OA) blood flow parameters in the intracranial (IOA) and extracranial (EOA) segments of the OA with two-depth transcranial Doppler (TCD)). Based on the good results of the previous study, the study should be repeated in order to further validate the new method in more patients and to obtain additional insight with more measurements.

This single centre, observational comparative study shall investigate a new non-invasive ICP absolute value measurement method in patients presenting with TBI, ICH, or secondary edema after stroke or Subarachnoid Hemorrhage (SAH) compared to current standard invasive ICP monitoring methods.Suitable patients are to be recruited soonest after their referral or admission to the Department of Neurosurgery at the Kantonsspital Aarau. Measurement will be done either at the surgical Intensive Care Unit, Stroke Unit ("SIC") or Neurosurgical Intermediate Care Unit ("NCW"). All measurements will be performed on intubated and sedated patients with invasive ICP Monitoring trough an intraparenchymatous or intraventricular probe. In the same patient, several measurements will be allowed daily.

The non-invasive technique for measurement of ICP is based on simultaneously measuring of an ophthalmic artery (OA) blood flow parameters in the intracranial (IOA) and extracranial (EOA) segments of the OA with two-depth transorbital Doppler (TCD) measurements including mechanical head frame for fixation of ultrasonic transducer on the closed eye lid. ICP pressure will be measured non-invasively by using Vittamed 205® device. This device has CE marking since July 2014.

It is planned to recruit 25 patients and to collect 69 independent paired non-invasive and invasive ICP measurements during a 24 months period after study approval.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, age ≥ 18 years, admitted after TBI, ICH, secondary edema after stroke or SAH at the Departments of Neurosurgery or Neurology, Kantonsspital Aarau, Switzerland.
* Patients under sedation and ICP monitoring
* Informed consent obtained from the legally authorized representative prior initiation of the measurements.

Exclusion Criteria:

Age < 18 years at study entry.

* Patients with wounds, scars including the front orbital region.
* Perforating or penetrating mechanism of TBI
* Patients with orbital injury or abnormal blood flow in both Ophthalmic Arteries
* Patients with previous retina surgery
* Patients with previous cataract surgery
* Patients with any known ocular condition that may be worsened by sustained eye pressure in the opinion of the subject's ophthalmologist
* Patients with radiological signs of calcification or atheromatose plaques in the internal carotid artery detected by CT or angiography (performed prior and independently of the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients, age ≥ 18 years, after Traumatic Brain Injury, Intrcranial Hemorrhage, secondary edema after stroke or SAH
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Absolute intracranial pressure | 35 minutes per measurement
  absolute intracranial ICP, measured simultaneously with the non-invasive and the standard invasive method

OTHER OUTCOMES:
Safety outcome | during measurements
  Incidence of device related Adverse Events and Serious Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: jenny kienzler, Principal Investigator — Kantonsspital Aarau

IPD SHARING:
Plan to Share IPD: No